CLINICAL TRIAL: NCT05757479
Title: Efficacy and Safety of Saline Rinses Combined With Steroid-Eluting Stent Implant or Steroid Nasal Spray in Radiation-Related Sinusitis
Brief Title: Steroid-Eluting Stent Implant for the Treatment of Radiation-Related Sinusitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Zhongshan People's Hospital, Guangdong, China (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, professor & chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2022-sinusitis
Record Dates: First submitted 2023-02-13; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Radiation-Induced Mucositis
Keywords: Nasopharyngeal carcinoma; Radiation-related sinusitis; Steroid-eluting stent
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Nasal Lavage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroid-eluting stent implant (Experimental): Subjects randomized to the experimental group will receive steroid-eluting stent implantation in the affected sinus and saline rinses.
  Interventions: Procedure: Steroid-eluting stent implantation; Procedure: nasal saline rinses
- Nasal steroid spray (Active Comparator): Subjects randomized to the comparator group will receive nasal steroid spray and saline rinses.
  Interventions: Drug: Steroid nasal spray; Procedure: nasal saline rinses

INTERVENTIONS:
Procedure: Steroid-eluting stent implantation — The sinus cavity with inflammation receives one bioabsorbable steroid-eluting sinus stent.
  Arms: Steroid-eluting stent implant
Drug: Steroid nasal spray — 1 spray into each nostril once a day.
  Arms: Nasal steroid spray
Procedure: nasal saline rinses — The saltwater runs through nasal passages and drains out of the nostril.
  Other Names: Nasal irrigation

SUMMARY:
Sinusitis is one of the most common sequelae after radiotherapy among nasopharyngeal carcinoma patients. While local steroids have been shown to be effective in the management of patients with chronic rhinosinusitis, their role in treating radiation-related sinusitis is ambiguous. Poor adherence to nasal steroid spray often contributes to the failure of symptom relief. The aim of this study is to determine if steroids stents implantation into the sinuses could improve patient outcomes in radiation-related sinusitis.

DETAILED DESCRIPTION:
Investigators aim to assess the efficacy and safety of Steroid-eluting stents when implanted in sinus in patients with radiation-related sinusitis. This phase III randomized controlled study enrolled nasopharyngeal carcinoma patients who received radiotherapy and developed severe radiation-related sinusitis. Subjects were randomly assigned to receive steroid-eluting stents implantation or nasal steroid spray. All study patients also received saline rinses.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed nasopharyngeal carcinoma patients
* finished radical radiotherapy (≥66Gy) for at least 3 months
* tumor complete response
* received appropriate medical treatment for sinusitis during or after radiotherapy
* confirmed sinusitis according to European Position Paper on Rhinosinusitis and Nasal Polyps 2020
* SNOT-22 ≥ 20 and MRI Lund-Mackay score > 8
* 18-70 years old

Exclusion Criteria:

* anatomic variation resulted in occluded ostiomeatal complex
* Karnofsky score ≤ 70
* life-threatening medical conditions
* tumour residue or recurrence
* acute bacterial sinusitis or acute fungal sinusitis
* cystic fibrosis or primary ciliary dyskinesia
* dependence on prolonged corticosteroid therapy for comorbid conditions
* history of allergy to topical steroids
* pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-02-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Sino-Nasal Outcome Test Scores (SNOT-22) | Change from Baseline to Week 12
  The change in Sino-Nasal Outcome Test scores (SNOT-22) scores pre- and post-treatment between the two arms was measured. The Sino-Nasal Outcome Test asks subjects to rate how "bad" their rhinosinusitis is by using a 0-5 point scale with 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The SNOT includes 22 questions (symptoms and social/emotional consequences of rhinosinusitis), each of which are rated from 0 to 5 for a minimum score of 0 to maximum score of 110, with higher scores representing worse outcome.
Change in Lund-Mackay MRI score | Change from Baseline to Week 12
  Sinus MRI Lund-Mackay (LM) score (0-20). Higher score means more severe disease.

SECONDARY OUTCOMES:
Lund-Kennedy Scoring for Nasal Endoscopy | Change from Baseline to Week 12 and Week 24
  The Lund Kennedy scoring system for nasal endoscopy rates the severity of the sinusitis based on the endoscopic appearance of the nasal mucosa. Edema, secretions and the presence of polyps are rated from 0-2, for a total maximum score of 6 per each side of the nose. Higher scores represent more severe disease.
Change in Sino-Nasal Outcome Test Scores (SNOT-22) | Change from Baseline to Week 4 and Week 24
  The change in Sino-Nasal Outcome Test scores (SNOT-22) scores pre- and post-treatment between the two arms was measured. The Sino-Nasal Outcome Test asks subjects to rate how "bad" their rhinosinusitis is by using a 0-5 point scale with 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The SNOT includes 22 questions (symptoms and social/emotional consequences of rhinosinusitis), each of which are rated from 0 to 5 for a minimum score of 0 to maximum score of 110, with higher scores representing worse outcome.
Change in Quality of life using The European Organization for Research and Treatment of Cancer core quality of life questionnaire（EORTC QLQ-30） | Change from Baseline to Week 12 and Week 24
  Comparison of quality of life using questionnaires EORTC QLQ-30. All EORTC QLQ-C30 scale scores range from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptom-atology.
Change in Quality of life using questionnaires EORTC QLQ-Head&Neck35 (HN35) | Change from Baseline to Week 12 and Week 24
  Comparison of quality of life using questionnaires HN35. HN35 score ranges from zero to 100. A high score for a functional or global scale represents a relatively high/healthy level of functioning or global quality of life, whereas a high score for a symptom scale represents the presence of a symptom or problem(s).
Rescue medication | Week 12 and Week 24
  Rescue medication use of corticosteroids and antibiotics. Specifically, total usage over six month period.
The effective rate | Week 12 and Week 24
  Cure: the symptoms disappeared, sinus ostium open, and the sinus mucosa was epithelialized without purulent secretions.
  Improved: the symptoms were significantly improved. Endoscopic examination showed edema, hypertrophy or granulation tissue formation in some areas of sinus mucosa, and a small amount of purulent secretions.
  Ineffective: the symptoms were not improved. Endoscopic examination showed stenosis or atresia of the sinus ostium, formation of polyps or purulent secretions.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD, PhD, Study Chair — Sun Yat-sen University
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China